CLINICAL TRIAL: NCT02224534
Title: High PlatElet Inhibition With TicAgrelor to Improve Left Ventricular RemodeLING in Patients With ST-segment ElevAtion Myocardial Infarction: the HEALING-AMI Trial.
Brief Title: Ticagrelor Versus Clopidogrel in Left Ventricular Remodeling After ST-segment Elevation Myocardial Infarction
Acronym: HEALING-AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gyeongsang National University Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Chungnam National University Hospital (Other); Pusan National University Yangsan Hospital (Other); National University Heart Centre, Singapore (Other); Ulsan University Hospital (Other); Kyungpook National University Hospital (Other); Samsung Changwon Hospital (Other); Kyunghee University Medical Center (Other); Chungbuk National University Hospital (Other); Chonnam National University Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yongwhi Park, MD.,PhD., Gyeongsang National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5130C00138
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST elevation myocardial infarction.; Ticagrelor; Left ventricular remodeling; Platelet reactivity
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Remodeling | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor and Clopidogrel. (Experimental): The patients assigned to the TICA group have loading dose of ticagrelor 180 mg just after the randomization, and then ticagrelor 90 mg twice daily during the study period. All patients also have aspirin 300 mg as a loading dose and 100 mg once daily as a maintenance dose.
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): The patients assigned to the CLPD group have loading dose of clopidogrel 600 mg just after the randomization, and then clopidogrel 75 mg daily should be maintained during the study period. All patients also have aspirin 300 mg as a loading dose and 100 mg once daily as a maintenance dose.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 180 mg as a loading dose and 90 mg twice daily as a maintenance dose
  Other Names: Brillinta
  Arms: Ticagrelor and Clopidogrel.
Drug: Clopidogrel — Clopidogrel 600 mg as a loading dose and 75 mg once daily as a maintenance dose.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The purpose of the study is to evaluate the novel role of ticagrelor to improve long-term LV remodeling following ST-segment elevation myocardial infarction.

DETAILED DESCRIPTION:
The investigators designed the HEALING-AMI study to compare the influence of ticagrelor (180 mg loading and 90 mg twice daily maintenance) vs. clopidogrel (600 mg loading and 75 mg daily maintenance) on long-term left ventricular (LV) remodeling measured by 3D echocardiography in STEMI patients undergoing primary PCI.

The primary objective of the HEALING-AMI study is to demonstrate the novel role of long-term ticagrelor therapy in reducing the risk of LV remodeling,. The secondary objectives are to reveal the cross-talk between platelet and inflammatory process in ST-segment elevation myocardial infarction (STEMI) patients. Moreover, this study will determine whether the high platelet inhibition by ticagrelor culminate the protection of infarcted myocardium.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* First-time onset STEMI patients uneventfully treated with primary PCI within 12 hours of onset of symptom.
* Infarct-related artery with TIMI 0, 1, or 2 grade flow at the time of initial diagnostic angiography (before wire passage).
* proximal or mid-portion lesion of epicardial coronary artery.

Exclusion Criteria:

* Previous history of myocardial infarction.
* Left bundle branch block on ECG at the time of screening.
* Cardiogenic shock at the time of randomization.
* Refractory ventricular arrhythmias or atrial fibrillation.
* New York Heart Association class IV congestive heart failure.
* Severe or malignant hypertension (SBP> 180 and/or DBP> 120 mmHg).
* Fibrinolytic therapy.
* History of hemorrhagic stroke.
* Intracranial neoplasm, arteriovenous malformation, or aneurysm.
* Ischemic stroke within 3 months prior to screening.
* Platelet count < 100,000/mm3 or hemoglobin < 10 g/dL.
* A need for oral anticoagulation therapy that cannot be safely discontinued for the duration of the study.
* Women who are known to be pregnant, have given birth within the past 90 days, or are breast-feeding.
* Unable to cooperate with protocol requirements and follow-up procedures.
* A history of P2Y12 receptor inhibitor pretreatment (at least prior 1 month).
* An increased risk of bradycardia.
* Concomitant therapy with a strong cytochrome P-450 3A inhibitor or inducer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
LV remodeling index (%) | Interval change between baseline and 6 months after the index events
  Real time 3D-echocardiography data sets will be analyzed with available 4D-LV Analysis software (e.g. TomTec Imaging Systems, Unterschleisheim, Germany) in the core lab.
  Left ventricular (LV) remodeling index: a relative change in LV end-diastolic volume (LVEDV) seen at 6-month follow-up compared with the baseline during admission.
NT-proBNP level at 6 months | 6 months after the index events

SECONDARY OUTCOMES:
Absolute change of LVESVI, LVEDVI and LVEF | Interval change between baseline and 6 months after the index events
Prevalence of adverse LV remodeling | Interval change between baseline and 6 months after the index events
  Adverse LV remodeling: a relative > 20% increase in LVEDV seen at 6-month follow-up compared with the baseline during admission.
Level of platelet reactivity | At the time of PCI, 3 days and 1 month after the events
  Measured by VerifyNow P2Y12 assay

OTHER OUTCOMES:
Post-PCI angiographic perfusion indicators: TIMI flow grade, myocardial blush grade, corrected TIMI frame count | Just after primary PCI
EKG change: ST-segment elevation resolution (%), complete ST-segment resolution | Baseline, 60 minutes after the PCI.
  complete ST-segment resolution: ST-segment resolution ≥70%
Level of hs-CRP | At the time of PCI, 1 month and 6 months after the events
Bleeding events based on BARC or PLATO definition | 6 months after the events
  BARC definition for bleeding is defined as type 1, 2, 3 (3a, 3b and 3c), 4, and 5 (5a and 5b), according to the Bleeding Academic Research Consortium classification.
  * Type 1 (nuisance or superficial bleeding).
  * Type 2 (internal bleeding).
  * Type 3a (TIMI minor bleeding).
  * Type 3b (TIMI major bleeding).
  * Type 3c (life threatening bleeding).
  * Type 4 (CABG-related bleeding).
  * Type 5a (probable fatal bleeding).
  * Type 5b (definite fatal bleeding). Bleeding events pertaining to type 1 to 3a are considered as minor bleeding and those pertaining to type 3b to 5b as major bleeding.
  PLATO definition for bleeding
  * Major life-threatening bleeding.
  * Other major bleeding.
  * Minor bleeding.
  The case report form (CRF) collects the event history of bleeding during admission and at 1 month and 6 months. Occurrences of major, minor, and combined major and minor bleeding events will be compared between groups.
Cardiac MRI (Substudy): LV remodeling index | Three days and 6 months after the events
  Measured at A*STAR-NUS Clinical Imaging Research Centre, Singapore
Level of inflammatory markers (Substudy) | During hospitalization and at 1 month after the events

CONTACTS AND LOCATIONS:
Overall Officials: Yongwhi Park, MD., PhD., Principal Investigator — Gyeongsang National University Hospital; Young-Hoon Jeong, MD.,PhD., Principal Investigator — Gyeongsan National University Hospital
Locations (12):
- Chinese PLA General Hospital, Beijing, China
- National University Heart Centre, Singapore, Singapore
- South Korea (10):
  - Chonnam National University Hospital, Gwangju, CHONRANAM-Do
  - Seoul National University Bundang Hospital, Bundang, Gyeongki-do
  - Changwon Samsung Medical Center, Changwon
  - Chungbuk National University Hospital, Chungju
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Gyeongsang National University Hospital, Korea
  - Kyung Hee University Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park Y, Koh JS, Lee JH, Park JH, Shin ES, Oh JH, Chun W, Lee SY, Bae JW, Kim JS, Kim W, Suh JW, Yang DH, Hong YJ, Chan MY, Kang MG, Park HW, Hwang SJ, Hwang JY, Ahn JH, Choi SW, Jeong YH; HEALING-AMI Investigators. Effect of Ticagrelor on Left Ventricular Remodeling in Patients With ST-Segment Elevation Myocardial Infarction (HEALING-AMI). JACC Cardiovasc Interv. 2020 Oct 12;13(19):2220-2234. doi: 10.1016/j.jcin.2020.08.007. PMID 33032710
- [Derived] Park Y, Choi SW, Oh JH, Shin ES, Lee SY, Kim J, Kim W, Suh JW, Yang DH, Hong YJ, Chan MY, Koh JS, Hwang JY, Park JH, Jeong YH; HEALING-AMI Trial Investigators. Rationale and Design of the High Platelet Inhibition with Ticagrelor to Improve Left Ventricular Remodeling in Patients with ST-Segment Elevation Myocardial Infarction (HEALING-AMI) Trial. Korean Circ J. 2019 Jul;49(7):586-599. doi: 10.4070/kcj.2018.0415. Epub 2019 Mar 22. PMID 31074220